CLINICAL TRIAL: NCT00944489
Title: Hypertension and Health-Related Quality of Life Adherence: Cross- Sectional Observational Study in Ambulatory Patients
Brief Title: To Assess Adherence to the Treatment and Quality of Life in Patients With Hypertension
Acronym: ADHERENCE
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: MC MD, AstraZeneca
Other Study IDs: NIS-CAR-ATA-2009/1
Record Dates: First submitted 2009-07-17; First posted 2009-07-23 (Estimated); Last update posted 2010-12-07 (Estimated); Status verified 2010-12

CONDITIONS: Hypertension
Keywords: Hypertension; Health-Related Quality of Life Adherence to the antihypertension treatment; Ambulatory Patients; MINICHAL score; Treatment Adherence Scale (MMAS); Quality of life; Adherence to treatment
MeSH Terms: conditions — Hypertension; Treatment Adherence and Compliance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients with diagnosis of essential hypertension under the criteria established by the Joint National Committee VII (9) and those patients under pharmacological treatment with the same therapeutic regime during at least the last 6 months.

SUMMARY:
The main goal of this study is to achieve a deeper knowledge of the adherence to antihypertensive drug treatment and to evaluate the quality of life in this population. This work has the following goals: primary objective is to assess the antihypertensive treatment adherence in patients with essential hypertension on treatment for more than 6 months.

The secondary objectives include the assessment of quality of life, identification of associated factors that affect adherence, knowledge of drugs used and comparison of levels of adherence according to the different drug regimes

Two questionnaires shall be prepared The first questionnaire shall be anonymously completed by the patient willing to participate. It is divided into two parts:

1. Treatment Adherence Scale (MMAS): this survey is made up of 4 questions having YES/No answers and it grants 1 point per every "NO" answer, and zero points to every "YES" answer.
2. The second part is the health-related quality of life Questionnaire (MINICHAL). The questions refer to the "last 7 days" with 4 possible answer options: 0 (no, absolutely not), 1 (yes, sometimes), 2 (yes, frequently) and 3 (yes, a lot). It is made up of 16 items, 10 correspond to the "State of Mind" dimension and 6 to the "Body-related Symptoms," also described as "Physical symptoms".

The second questionnaire shall be completed by the intervening physician as regards patients that attend medical visits, and who have answered the anonymous questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosis of essential hypertension under the criteria established by the Joint National Committee VII (9) and those patients under pharmacological treatment with the same therapeutic regime during at le

Exclusion Criteria:

* Patients with secondary HBP
* Pregnant women or nursing mothers
* Patients with acute illnesses or having a definite psychiatric diagnosis, as well as those patients who are unable to completed

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: clinic and private practice
Sampling Method: Probability Sample
Enrollment: 1150 (Actual)
Dates: Start 2009-08; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
First questionnaires for patient:Treatment Adherence Scale, and the health-related quality of life Questionnaire .the intervening physician completed second questionnaire with all about the non and pharmacology treatment | 3-6 months

SECONDARY OUTCOMES:
Assess quality of life in patients in this cohort. | 3-6 months
Identify associated factors that may alter adherence to antihypertensive treatment. | 3-6 months
Know pharmacological groups used for this pathology and compare treatment adherence level according to the different therapeutic regimes used | 3-6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Buenos Aires, Argentina